CLINICAL TRIAL: NCT02478684
Title: The Effects of Delayed Cord Clamping on Postnatal Circulatory Status in Preterm Neonates
Brief Title: Delayed Cord Clamping in Preterm Neonates
Acronym: DCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1411015633
Record Dates: First submitted 2015-06-11; First posted 2015-06-23 (Estimated); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Premature Birth of Newborn; Infant, Very Low Birth Weight; Delayed Separation of Umbilical Cord; Placental Transfusion
Keywords: delayed cord clamping; premature infants; randomized study; hematocrit
MeSH Terms: conditions — Premature Birth; Fetofetal Transfusion | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30 seconds of DCC (Active Comparator): 30 Seconds of placental blood transfusion
  Interventions: Other: 30 Seconds of placental blood transfusion
- 60 seconds DCC (Active Comparator): 60 Seconds of placental blood transfusion
  Interventions: Other: 60 Seconds of placental blood transfusion

INTERVENTIONS:
Other: 30 Seconds of placental blood transfusion — By delaying clamping of the cord blood for 30 seconds, blood will be allowed to move from the placenta to the premature infant
  Other Names: 30 Seconds of Delayed Cord Clamping
  Arms: 30 seconds of DCC
Other: 60 Seconds of placental blood transfusion — By delaying clamping of the cord blood for 60 seconds, blood will be allowed to move from the placenta to the premature infant
  Other Names: 60 Seconds of Delayed Cord Clamping
  Arms: 60 seconds DCC

SUMMARY:
Delayed cord clamping (DCC) from 30 to 60 seconds allows blood to continue to flow from the placenta through the umbilical cord to the infant, thus resulting in a placental transfusion. This transfusion may improve circulating volume at birth leading to a smoother postnatal transition and overall improved outcome for preterm infants. The average blood volume delivered with DCC up to 90 seconds in preterm infants has been estimated to be about 12 ml per kg with vaginal deliveries resulting in slightly higher transfusions compared to cesarean deliveries. Several several short-term benefits have been described including a reduction in the need for blood transfusions as well as a possible reduction in intraventricular hemorrhage and necrotizing enterocolitis. All mothers with threatened preterm delivery between 28 and 34 6/7 weeks will be approached for the study. Following consent, the infant will be randomly assigned to either a 30 or 60 second delay in cord clamping in the delivery room. If the infant is not breathing by 30 seconds, the cord will be clamped and the infant moved to a resuscitation area. The primary outcome is a 3 percent difference in the hematocrit at one hour (routinely obtained on all babies). With approximately 75 neonates in each group (30 and 60 second DCC), there is 80% power to detect a difference in the mean hematocrit of 3% using a two-sample t-test with a 0.05 two-sided significance level.

DETAILED DESCRIPTION:
Placental transfusion at birth is thought to have immediate, short-term and long-term benefits for the neonate. Delaying cord clamping is thought to allow for a smoother postnatal transition as the necessary cardiopulmonary changes take place specifically when the infant establishes spontaneous respirations and/or experimentally when mechanical ventilation is initiated. By allowing the infant to establish respirations, the pulmonary vascular bed is able to relax prior to the removal of the low-resistance placental vascular bed, thus avoiding a reflexive bradycardia. A 2012 Cochrane review of DCC in preterm infants has suggested several short-term benefits including a reduction in the need for blood transfusions as well as a possible reduction in intraventricular hemorrhage and necrotizing enterocolitis. The American College of Obstetrics and Gynecology (ACOG) published a committee opinion in December of 2012 stating that current evidence supports delayed cord clamping in preterm infants. They go on to support that DCC up to 30-60 seconds has been shown to improve transitional circulation, decreased the need for blood transfusion, and may even reduce the incidence of intraventricular hemorrhage. The primary objective of this study is to determine if delayed cord clamping up to 60 seconds leads to an improved postnatal transition as demonstrated by higher initial hematocrit at 30 minutes in preterm neonates born between 28 and 34+6/7 weeks gestation. The investigators will determine whether there is a significant difference in this primary outcome with delays of 30 seconds versus 60 seconds. A secondary objective will be to determine the effect of DCC on additional measures such as Apgar scores, initial heart rate, initial temperature, blood pressure measures, fluid resuscitation and/or the need for pressors, peak bilirubin, and days on phototherapy.

Inclusion Criteria: Preterm infants born between 28 and 34+6/7 weeks gestation. Exclusion Criteria: Infant with suspected placental abruption, bleeding from placenta previa, terminal bradycardia, cord prolapse, meconium, or any major congenital anomalies.

All mothers with threatened preterm delivery between 28 and 34 6/7 weeks will be approached for the study. If consent is obtained, the infant will be randomly assigned to either a 30 or 60 second delay of cord clamping in the delivery room. All delivery room staff will be notified of the assignment prior to the delivery. The Neonatal Intensive Care Unit (NICU) staff will be present at each delivery, including a NICU Fellow, a NICU nurse, and/or an neonatal nurse practitioner or pediatric resident. In the case of a C-Section, the NICU fellow will be in sterile gown and gloves in order to assess the infant on the sterile field. The timer will start immediately following delivery of the entire infant. In the case of a vaginal delivery the infant will be placed between the mother's legs or on the mother's abdomen in the case of a cesarean section. The fellow will evaluate the infant to assess onset of respirations while stimulating and covering the infant in a plastic wrap. If the infant has good tone and sustained breathing, the umbilical cord will continue to be unclamped though a maximum of 60 seconds. If the infant has not begun to establish respirations at 30 seconds, the cord will be clamped and the infant will be transferred to the radiant warmer regardless of their original assignment.

The primary outcome is a 3 percent difference in the hematocrit at one hour (routinely obtained on all babies). With approximately 75 neonates in each group (30 and 60 second DCC), there is 80% power to detect a difference in the mean hematocrit of 3% using a two-sample t-test with a 0.05 two-sided significance level.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants between 28 and 34 6/7 weeks
* Parents have given informed consent

Exclusion Criteria:

* Suspected placental abruption
* Bleeding from placenta previa
* Terminal bradycardia
* Cord prolapse
* Meconium
* Any major congenital anomalies

Ages: 28 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2015-07; Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Measurement of Hematocrit at one hour of life | 18 months
  There should be a 3% difference between the 30 second and 60 second arms.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Perlman, MB Ch B, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kugelman A, Borenstein-Levin L, Riskin A, Chistyakov I, Ohel G, Gonen R, Bader D. Immediate versus delayed umbilical cord clamping in premature neonates born < 35 weeks: a prospective, randomized, controlled study. Am J Perinatol. 2007 May;24(5):307-15. doi: 10.1055/s-2007-981434. Epub 2007 May 21. PMID 17516307
- [Background] Mercer JS, McGrath MM, Hensman A, Silver H, Oh W. Immediate and delayed cord clamping in infants born between 24 and 32 weeks: a pilot randomized controlled trial. J Perinatol. 2003 Sep;23(6):466-72. doi: 10.1038/sj.jp.7210970. PMID 13679933
- [Background] Mercer JS, Vohr BR, McGrath MM, Padbury JF, Wallach M, Oh W. Delayed cord clamping in very preterm infants reduces the incidence of intraventricular hemorrhage and late-onset sepsis: a randomized, controlled trial. Pediatrics. 2006 Apr;117(4):1235-42. doi: 10.1542/peds.2005-1706. PMID 16585320
- [Background] Oh W, Fanaroff AA, Carlo WA, Donovan EF, McDonald SA, Poole WK; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Effects of delayed cord clamping in very-low-birth-weight infants. J Perinatol. 2011 Apr;31 Suppl 1(Suppl 1):S68-71. doi: 10.1038/jp.2010.186. PMID 21448208
- [Background] Rabe H, Wacker A, Hulskamp G, Hornig-Franz I, Schulze-Everding A, Harms E, Cirkel U, Louwen F, Witteler R, Schneider HP. A randomised controlled trial of delayed cord clamping in very low birth weight preterm infants. Eur J Pediatr. 2000 Oct;159(10):775-7. doi: 10.1007/pl00008345. PMID 11039135
- [Background] Strauss RG, Mock DM, Johnson KJ, Cress GA, Burmeister LF, Zimmerman MB, Bell EF, Rijhsinghani A. A randomized clinical trial comparing immediate versus delayed clamping of the umbilical cord in preterm infants: short-term clinical and laboratory endpoints. Transfusion. 2008 Apr;48(4):658-65. doi: 10.1111/j.1537-2995.2007.01589.x. Epub 2008 Jan 10. PMID 18194383
- [Background] Aladangady N, McHugh S, Aitchison TC, Wardrop CA, Holland BM. Infants' blood volume in a controlled trial of placental transfusion at preterm delivery. Pediatrics. 2006 Jan;117(1):93-8. doi: 10.1542/peds.2004-1773. PMID 16396865
- [Background] Baenziger O, Stolkin F, Keel M, von Siebenthal K, Fauchere JC, Das Kundu S, Dietz V, Bucher HU, Wolf M. The influence of the timing of cord clamping on postnatal cerebral oxygenation in preterm neonates: a randomized, controlled trial. Pediatrics. 2007 Mar;119(3):455-9. doi: 10.1542/peds.2006-2725. PMID 17332197
- [Background] Hofmeyr GJ, Bolton KD, Bowen DC, Govan JJ. Periventricular/intraventricular haemorrhage and umbilical cord clamping. Findings and hypothesis. S Afr Med J. 1988 Jan 23;73(2):104-6. PMID 3340910
- [Background] Hofmeyr GJ, Gobetz L, Bex PJ, Van der Griendt M, Nikodem C, Skapinker R, Delahunt T. Periventricular/intraventricular hemorrhage following early and delayed umbilical cord clamping. A randomized controlled trial. Online J Curr Clin Trials. 1993 Dec 29;Doc No 110:[2002 words; 26 paragraphs]. PMID 8305996
- [Background] Kinmond S, Aitchison TC, Holland BM, Jones JG, Turner TL, Wardrop CA. Umbilical cord clamping and preterm infants: a randomised trial. BMJ. 1993 Jan 16;306(6871):172-5. doi: 10.1136/bmj.306.6871.172. PMID 8443480
- [Background] McDonnell M, Henderson-Smart DJ. Delayed umbilical cord clamping in preterm infants: a feasibility study. J Paediatr Child Health. 1997 Aug;33(4):308-10. doi: 10.1111/j.1440-1754.1997.tb01606.x. PMID 9323618
- [Result] Committee on Obstetric Practice, American College of Obstetricians and Gynecologists. Committee Opinion No.543: Timing of umbilical cord clamping after birth. Obstet Gynecol. 2012 Dec;120(6):1522-6. doi: 10.1097/01.AOG.0000423817.47165.48. PMID 23168790